CLINICAL TRIAL: NCT05539599
Title: Can Heart-lung-respiratory Muscles Ultrasound Evaluation Play a Role to Predict Weaning in Critically Ill Patients?
Brief Title: Comprehensive Ultrasound Evaluation as a Predictor of Weaning
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Fogagnolo, Principal investigator, Università degli Studi di Ferrara
Other Study IDs: WEAN_US
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Mechanical Ventilation Weaning; Weaning Failure
Keywords: weaning; MV critically ill patients; Ultrasound evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients will undergo a spontaneous breathing trial. Any extubation will be decided by an independent operator.
  Interventions: Diagnostic Test: Comprehensive evaluation

INTERVENTIONS:
Diagnostic Test: Comprehensive evaluation — Non-ultrasound parameters: Central venous pressure, hand-grip strength evaluation, P0.1, Maximal inspiratory pressure, Blood gas analysis ultrasound parameters: Diaphragmatic displacement, thickening fraction, TFmax, E/e', Triscuspidal annular Plane Systolic Excursion, Lung score

SUMMARY:
Several studies investigated the role of specific clinical predictors of weaning success, but it is determined by a combination of different aspects that can result in success or failure. Indeed, unresolved lung disease, cardiac dysfunction, loss of respiratory and core muscle strength can play a role in a failure weaning to mechanical ventilation (MV). The investigators hypothesized that a combined score that include heart, lung, and respiratory muscle ultrasound (US) evaluation could be able to predict the ability of weaning success. Furthermore, it will be described weather the days of MV before weaning trial may affect the relevance of each clinical variable evaluated.

DETAILED DESCRIPTION:
Critically ill patients undergone at least 48 hours of MV and ready to spontaneous breathing trial (SBT) will be included in the study. The spontaneous breathing trial is performed in pressure support ventilation with a clinician-set positive end expiratory pressure (PEEP) ≤ 5 cm H2O and FiO2< 40%. In addition to the parameters traditionally used for the evaluation of weaning (RSBI), the investigators will perform ultrasound evaluation of diaphragm, lung parenchyma, cardiac function, and the strength of the hand grip.

Investigators will evaluate the diaphragmatic parameters (thickening fraction,TF, and diaphragmatic displacement, DD) and TFmax (TF during forced breathing /TF during tidal respiration) to identify the inspiratory reserve. Weaning success is considered as liberation from MV within 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 90 years
* Mechanical ventilation> 48 h
* Reason for ICU admission: medical / surgical / trauma

Exclusion Criteria:

* age under 18
* diagnosis of neuromuscular disease
* tracheostomy
* terminal extubation
* pregnancy in progress -
* previous paralysis of the diaphragm or of a hemidiaphragm
* use of neuromuscular blocking drugs in continuous infusion in the 48 hours preceding the weaning attempt.
* Refusal to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated patients
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Assessing the prognostic value of a combined score in predicting weaning success | 72 hours
  We hypothesized that a combined score that include heart, lung, and respiratory muscle ultrasound (US) evaluation could be able to predict the ability of weaning success.

SECONDARY OUTCOMES:
Interaction between days of mechanical ventilator and determinant of weaning success | 28 days
  We will assess the interaction between days of mechanical ventilation and the prognostic value of Central venous pressure, hand-grip strength evaluation, P0.1, Maximal inspiratory pressure, Blood gas analysis, Diaphragmatic displacement, thickening fraction, TFmax, E/e', Triscuspidal annular Plane Systolic Excursion, Lung score in predicting weaning success

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università di Ferrara, Ferrara
  - Università di Siena, Siena